CLINICAL TRIAL: NCT02629731
Title: Quantitative Prescription of Foot Orthoses: A Dose-Response Study of Kinematics in Patients With Foot and Ankle Pain Using Biplane Fluoroscopy
Brief Title: Orthotic Dose Response Study
Acronym: ODRS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Collaborators: University of Washington (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Factorial | Masking: None | Purpose: Basic Science
Other Study IDs: O2008-R
Record Dates: First submitted 2015-12-02; First posted 2015-12-14 (Estimated); Last update posted 2024-06-21 (Actual); Status verified 2024-06

CONDITIONS: Ankle Osteoarthritis; Flat Foot or Pes Planus
Keywords: foot; ankle; osteoarthritis; flat foot
MeSH Terms: conditions — Flatfoot; Osteoarthritis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- ankle OA (Experimental): inclusion criteria: 1) diagnosis of ankle OA or PTTD [non-control subjects only], 2) undergoing conservative care (i.e., prescribed a foot orthosis) and deemed not to be a surgical candidate, 3) between 18 and 80 years of age, and 4) ambulatory (able to walk at least 15 m) with the primary impediment to pain-free ambulation being ankle OA or PTTD
  Interventions: Device: custom orthoses with varying degrees of hindfoot posting
- flat foot (Experimental): inclusion criteria: 1) diagnosis of flat foot, 2) undergoing conservative care (i.e., prescribed a foot orthosis) and deemed not to be a surgical candidate, 3) between 18 and 80 years of age, and 4) ambulatory (able to walk at least 15 m)
  Interventions: Device: custom orthoses with varying degrees of hindfoot posting
- control (No Intervention): inclusion criteria: 1) between 18 and 80 years of age, and 2) ambulatory (able to walk at least 15 m)

INTERVENTIONS:
Device: custom orthoses with varying degrees of hindfoot posting — The base orthotic design will be altered for one foot (most symptomatic in the case of patients or randomly chosen for controls) to give variations from 5-degree lateral hindfoot posting to 10-degree medial in 2.5-degree increments.
  Arms: ankle OA; flat foot

SUMMARY:
This study will investigate the effect of foot orthoses on two common conditions (ankle osteoarthritis and symptomatic adult onset flat feet) by using a custom biplane X-ray system the group has developed to very accurately and precisely quantify foot bone motion. The investigators will vary the design of the orthoses and subjects will be examined to find out which are most effective at improving function.

DETAILED DESCRIPTION:
The aim with this proposal is to better understand how in-shoe foot orthoses achieve improvements in foot and ankle function for people with ankle osteoarthritis (OA) and/or adult acquired flatfoot resulting from posterior tibial tendon dysfunction (PTTD). The investigators also aim to be able to predict what the optimal, personalized orthotic device is for each patient is. These are common, painful, and often highly debilitating conditions, with ankle OA estimated to affect around 6% of the adult population and adult acquired flat foot around 3.3% percent of females. It has been shown that foot orthoses can be an effective conservative intervention for these conditions, and can help to postpone or negate surgery. However, for a significant proportion of patients foot orthoses are unsuccessful, and there is evidence that this may be a result of significant inter-individual variability in joint movement and loading response to the intervention. This may be due to a number of factors, including foot bone shape, muscle strength, and/or joint range of motion. In addition, the design of foot orthoses is often inconsistent between suppliers, largely because of the manual approach that is used to design and manufacture them. A further complicating factor is that prescriptions for foot orthoses are often vaguely written. Improving the investigators' understanding of different foot and ankle responses to variation in foot orthotic design is essential if the investigators are to improve how these devices function at the level of the individual patient. To measure how the individual bones of the foot move using traditional techniques is, however, very difficult. Such methods rely on skin-mounted markers that are tracked in space to determine foot and ankle kinematics. However the size and position of the foot and ankle bones means that it is not possible to measure them all of them individually. Moreover, the movement between the skin and the underlying bones, known as soft tissue artifact, introduces significant errors into the measurements. This is further complicated by the need to wear shoes for orthoses to function properly. The group has developed a biplane fluoroscopy system that is tailored to address the unique issues of measuring foot kinematics. This system has the additional advantage of being able to measure the effects of foot orthotics in unmodified shoes. To achieve the objective of understanding and being able to predict the effects of orthoses, the specific aims are:

* [1]: To collect, via biplane fluoroscopy, kinematic data describing the effect of varying the angle of hindfoot posting in foot orthotics. These data will be obtained from 90 participants: 30 with ankle OA; 30 with symptomatic PTTD; and 30 healthy controls.
* [2]: Using the data from SA1, carry out a regression analysis to identify factors obtained from biplane fluoroscopy and clinical exam that significantly influence an individual's response (i.e., hindfoot kinematics) to the orthotic intervention. These factors include: foot type, bone geometry, static foot posture, joint axis location, range of motion, and muscle strength.
* [3]: Using the data from SA1, generate a musculoskeletal model of the foot that allows detailed analysis of the muscles and ligaments controlling ankle movement. This will be developed in the OpenSim modeling platform and made freely available upon project completion.
* [4]: To compare the kinematic responses to orthotic devices prescribed using standard methods and those prescribed using algorithms and insight from SA2 and SA3 in a separate group of participants. Biplane fluoroscopy will be used to collect kinematic data from 10 patients with ankle OA and 10 with PTTD to compare the performance of the three pairs (one traditional, one from SA2 and one from SA3) of orthotics. This data will also be used to validate the predictions resulting from SA2 and SA3. This proposed research project will improve the investigators' understanding of how foot orthotics work and will help us to prescribe more effective devices to patients. This will benefit the large number of people in the population with ankle osteoarthritis and adult acquired flat foot.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of ankle OA or PTTD [non-control subjects only]
* undergoing conservative care (i.e., prescribed a foot orthosis) and deemed not to be a surgical candidate
* between 18 and 80 years of age
* ambulatory (able to walk at least 15 m) with the primary impediment to pain-free ambulation being ankle OA or PTTD

Exclusion Criteria:

Exclusion criteria for all subjects include:

* recent (<1 year) surgical, neurological, metabolic or lower limb musculoskeletal problem that might impair the ambulation measures in the study, such as severe knee or hip osteoarthritis
* rheumatoid arthritis or other inflammatory disease
* foot ulceration or partial foot amputation
* inadequate cognitive or language function to consent or to participate
* lack of a telephone number or stable mailing address

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2016-07-01 (Actual); Primary Completion 2022-05-31 (Actual); Study Completion 2023-12-29 (Actual)

PRIMARY OUTCOMES:
peak hindfoot eversion | immediate
  In the proposed experiments, normal and pathological subjects will be studied while they walk with seven different designs of in-shoe orthoses in standardized footwear. Subjecting individuals to different "doses" of orthotic correction will generate "dose-response" curves (i.e., the kinematic variables) that will then be associated with patient-specific characteristics.
peak tibial rotation in degrees | immediate
  In the proposed experiments, normal and pathological subjects will be studied while they walk with seven different designs of in-shoe orthoses in standardized footwear. Subjecting individuals to different "doses" of orthotic correction will generate "dose-response" curves (i.e., the kinematic variables) that will then be associated with patient-specific characteristics.

CONTACTS AND LOCATIONS:
Overall Officials: William R. Ledoux, PhD, Principal Investigator — VA Puget Sound Health Care System Seattle Division, Seattle, WA
Locations (2):
- United States (2):
  - VA Puget Sound Health Care System Seattle Division, Seattle, WA, Seattle, Washington
  - University of Washington, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No